CLINICAL TRIAL: NCT07342400
Title: A Multi-center, Prospective Clinical Study to Assess Histological Changes From Treatment of Poly L-lactic Acid Biostimulator on Women at Various Menopausal Stages
Brief Title: A Clinical Study to Assess Histological Changes From Treatment of Poly L-lactic Acid Biostimulator on Women at Various Menopausal Stages
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.049
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Cheek Wrinkles; Menopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): All subjects have moderate-to-severe cheek wrinkles and will be treated with Sculptra three times, 4 weeks apart.
  Interventions: Device: Sculptra®

INTERVENTIONS:
Device: Sculptra® — Biostimulator

SUMMARY:
To assess protein expression stimulated by poly L-lactic acid (PLLA) via punch biopsy at each follow-up visits compared to Baseline.

DETAILED DESCRIPTION:
This is a randomized, prospective study. This study will enroll approximately 40 subjects across two sites. All subjects have moderate-to-severe cheek wrinkles on both cheeks.

Eligible subjects will first receive punch biopsy on one pre-auricular side according to a pre-determined randomization, followed by a first Sculptra treatment on both cheeks starting at the pre-auricular areas first at Baseline visit. Subjects will receive second Sculptra treatment at Week 4, and an optional third treatment at Week 8. At 12 weeks since last Sculptra treatment, half of the subjects will receive a second punch biopsy on the other pre-auricular side (per randomization). Subjects will have a follow up visit at 24 weeks since last Sculptra treatment. At 36 weeks since last Sculptra treatment, the remaining half will receive a second punch biopsy on the other pre-auricular side (per randomization).

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with symmetrical, moderate-to-severe cheek wrinkles on each side of the face as assessed via the Galderma Cheek Wrinkles Scale.
* Subject with intent to undergo correction of cheek augmentation or contour deficiencies
* Subjects willing to have a 3-mm punch biopsy on each preauricular side
* Subjects willing to maintain the current lifestyle, daily routine (e.g., diet, exercise, sleep, etc.), and a stable Body Mass Index (BMI, ± 5 kg/m2) throughout the study
* Ability of giving consent for participation in the study.
* Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

* Subjects with asymmetrical severity or unidentical cheek wrinkle score between 2 sides of the cheek.
* Subjects with a history of allergy or hypersensitivity to any ingredient of the treatment products.
* Previous tissue-augmenting therapy, contouring, or revitalization treatment in the face, except lips.
* Previous treatment/procedure in the face in the previous 6 months that, in the Investigator's opinion, would interfere with the study injections and/or study assessments or exposed the study subject to undue risk by study participation, or planning to undergo any of these procedures affecting the treatment area at any time during the study.
* Subjects with any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Protein Expression | 12 weeks, 24 weeks, and 36 weeks after Baseline
  Punch biopsies will be performed at the pre-auricular areas. Histology staining or immunohistochemistry will be performed on punch biopsy samples to evaluate targeted biomarkers compared to Baseline.

SECONDARY OUTCOMES:
Subject satisfaction using self-assessment questionnaire | 12 weeks, 24 weeks, and 36 weeks since final Sculptra treatment
  Subjects will be asked about their perception and satisfaction with the study treatments using a self-assessment questionnaire at visits after Baseline. The questionnaire will be a 5-point subject satisfaction questionnaire with the following responses: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami Dermatology & Laser Institute, Miami, Florida
  - Day Dermatology & Aesthetics, New York, New York

IPD SHARING:
Plan to Share IPD: No